CLINICAL TRIAL: NCT03468114
Title: The Safe Start Trial: a Cluster Randomised Controlled Trial for the Effect of a Food Hygiene Intervention on Infant Enteric Infections and Diarrhoeal Disease in Low-income Informal Settlements of Kisumu, Kenya.
Brief Title: The Safe Start Trial - Kisumu, Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Great Lakes University Kisumu (Other); University of Iowa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 14695
Record Dates: First submitted 2018-03-05; First posted 2018-03-16 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Enteric Infections; Diarrhea
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Masking Description: Outcome assessors are not informed of allocation but would likely infer this from the presence of highly visible domestic products that are part of the intervention. Lab technicians and data analysts are masked to allocation status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participant households will receive 4 visits by health extension workers delivering intervention
  Interventions: Behavioral: Safe Start
- Control (Active Comparator): Participant households will receive 4 visits by health extension workers delivering standard care
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Behavioral: Safe Start — Participant households will receive four visits over a 10 week period from health extension workers promoting safe food preparation, storage and feeding, and will be provided with products to support these practices (a bowl, spoon, cup, hand washing station, liquid soap dispenser).
  Arms: Intervention
Behavioral: Active Control — Participant households will receive 4 visits by health extension workers delivering standard care
  Arms: Control

SUMMARY:
This a cluster randomised controlled trial (cRCT) to evaluate the effect of a novel food hygiene intervention on infant health.

DETAILED DESCRIPTION:
Enteric infections remain a major threat to child health and development in many low and middle-income countries. Globally, diarrhoeal disease - a key health consequence of enteric infection - is ranked as the fourth leading cause of disability globally, after ischaemic heart disease, lower respiratory tract infections and strokes. Diarrhoeal disease persists as the second leading cause of child deaths in the world, and in sub-Saharan Africa is the leading cause of child deaths.

Public health efforts to address diarrhoeal disease have largely focused on improving access to safe drinking water and sanitation and promoting hand washing with soap to address faecal-oral routes of transmission. These interventions though may not effectively address all exposure pathways during early life, when young children are most susceptible to infection and the diarrhoeal disease burden is greatest. One potentially important exposure pathway is infant food which recent studies conducted in low income, high burden settings suggest may be highly contaminated and may be amenable to simple behaviour change interventions.

The Safe Start trial will evaluate the effect of a novel food hygiene intervention on infant health implemented in low income urban neighbourhoods of Kisumu, Kenya. The intervention is designed to target early childhood exposure to enteric pathogens through contaminated food and was developed through an earlier phase of formative behavioural and microbiological research. The intervention will target infant caregivers and be delivered through the Community Health Volunteer (CHV) health extension system. Four key behaviours will be addressed by the intervention:

1. Safe hand hygiene: handwashing with soap before infant food preparation and feeding
2. Safe food preparation: bringing all infant food to the boil before feeding, including when reheating
3. Safe storage of food: storing all infant food in sealed containers
4. Safe feeding: reserving specific feeding utensils for the infant and keeping these separate and clean

A cluster randomized controlled trial (cRCT) design will be used to evaluate the intervention with each CHV catchment area forming one cluster. The outcomes of interest for this study are as follows: (1) the prevalence of enteric infections among infants at 37 weeks of age (primary); (2) the longitudinal prevalence of diarrhoea between 22-37 weeks of age (primary); and (3) incidence of all-cause mortality between 22-37 weeks of age. Infants will be recruited on a rolling basis at 22 weeks of age (+/- 1 week), and data and/or samples collected at 3 points: baseline at 22 weeks of age (+/- 1 week); midline at 33 weeks of age (+/- 1 week); and endline at 37 weeks of age (+/- 1 week). Stool samples will be collected at baseline and endline and analysed for 23 genetic sequences indicating the presence of enteric pathogens known to cause childhood diarrhoea in low income, high burden settings.

ELIGIBILITY:
Inclusion Criteria:

* Infant is 21-23 weeks of age at enrolment
* Infant's mother residing within catchment of participating health extension worker at time of enrolment and intends to stay in current dwelling at least until infant reaches 37 weeks of age

Exclusion Criteria:

* Infant with any medical, psychiatric or social condition which, in the opinion of the research team, impedes the participant's ability to give informed consent

Ages: 21 Weeks to 23 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 880 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2019-05-09 (Actual); Study Completion 2019-06-22 (Actual)

PRIMARY OUTCOMES:
Enteric infection prevalence | At 37 weeks of age (+/- 1 week)
  Enteric infections are defined as the presence of enteric pathogens in stool as indicated by 1 or more of these 23 genetic sequences: Shigella/EIEC virulence plasmid, EAEC_aaic, EAEC_aata, EPEC_eae, EPEC_bfpa, ETEC_LT, ETEC_STp_STh, EHEC Escherichia coli 0157, Aeromonas, Vibrio cholerae, Campylobacter jejuni/C. coli, Clostridium difficile, and Salmonella enterica), Adenovirus 40/41, Adenovirus Hexon, Norovirus GI, Norovirus GII, and Rotavirus and broad reactive Cryptosporidium_18s, C. hominus, C. parvum, and Giardia assemblages A & B.
Diarrhoeal disease longitudinal prevalence | Between 22 and 37 weeks of age (+/- 1 week)
  Longitudinal prevalence is defined by days with diarrhoea during follow-up with diarrhoea defined according to WHO definition (3 or more loose or liquid stools passed within 24 hours)

OTHER OUTCOMES:
All-cause mortality incidence | Between 22 and 37 weeks of age (+/- 1 week)
  Deaths occurring during follow-up due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Cumming, MSc, Principal Investigator — London School of Hygiene and Tropical Medicine; Jane Mumma, PhD, Principal Investigator — Great Lakes University Kisumu
Locations (1):
- Great Lakes University Kisumu, Kisumu, Kenya

REFERENCES:
- [Derived] Baker KK, Mumma JAO, Simiyu S, Sewell D, Tsai K, Anderson JD, MacDougall A, Dreibelbis R, Cumming O. Environmental and behavioural exposure pathways associated with diarrhoea and enteric pathogen detection in 5-month-old, periurban Kenyan infants: a cross-sectional study. BMJ Open. 2022 Oct 31;12(10):e059878. doi: 10.1136/bmjopen-2021-059878. PMID 36316067
- [Derived] Mumma J, Simiyu S, Aseyo E, Anderson J, Czerniewska A, Allen E, Dreibelbis R, Baker KK, Cumming O. The Safe Start trial to assess the effect of an infant hygiene intervention on enteric infections and diarrhoea in low-income informal neighbourhoods of Kisumu, Kenya: a study protocol for a cluster randomized controlled trial. BMC Infect Dis. 2019 Dec 19;19(1):1066. doi: 10.1186/s12879-019-4657-0. PMID 31856747